CLINICAL TRIAL: NCT06129292
Title: The Effect of Emotional Freedom Technique on Breastfeeding in Women Experiencing Maternity Blues
Brief Title: The Effect of Emotional Freedom Technique on Breastfeeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Ayse Cuvadar, Assistant Professor, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TUTF_GOBAEK 2023/264
Record Dates: First submitted 2023-11-04; First posted 2023-11-13 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Breastfeeding
Keywords: Emotional Freedom Techniques; Breastfeeding; Maternity blues; Midwifery
MeSH Terms: conditions — Breast Feeding | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention (EFT) group (Experimental): Personal Information Form, Motherhood Blues Scale and Breastfeeding Self-Efficacy Scale will be applied for pre-test to women who meet our study criteria.
  To EFT Group; After the first tests are done, the 1st EFT session will be held, the 2nd EFT session will be held 10 days later, and the final tests will be done 10 days later. During this period, affirmations will be given depending on the need. Each session is planned to last an average of 45 minutes - 1 hour, and duration and affirmations will be arranged according to the woman's individual difficulties, perspective, support systems, past traumas and emotional blockages.
  Procedure 1: Preliminary tests will be carried out and then the 1st EFT session will be held.
  2nd Procedure: After 10 days, the first final tests will be performed and then the second EFT session will be held.
  Interventions: Behavioral: EFT group
- Control group (No Intervention): Personal information form, Motherhood Blues Scale and Breastfeeding Self-Efficacy Scale will be applied for pre-test to women who meet our study criteria. After 10 days, the motherhood blues scale and breastfeeding self-efficacy scale will be administered again for the final test.

INTERVENTIONS:
Behavioral: EFT group — Procedure 1: Preliminary tests will be carried out and then the 1st EFT session will be held.
  2nd Procedure: After 10 days, the first final tests will be performed and then the second EFT session will be held.
  Other Names: Control Group
  Arms: İntervention (EFT) group

SUMMARY:
This study was planned to determine the effect of the emotional liberation technique on breastfeeding in women experiencing motherhood sadness.

DETAILED DESCRIPTION:
Maternity blues is defined as a group of psychological and psychosomatic symptoms that generally affect women within 10-15 days after birth and are not considered a pathological condition. Emotional Freedom Techniques (EFT) is an evidence-based method that combines acupressure with elements from cognitive and exposure therapies. EFT has become widely used in medical and psychological treatment settings in recent years. It is also used as a self-help technique by millions of people every year.

For mothers experiencing motherhood blues, the opportunity to freely express and share their feelings can provide emotional relief. This can help reduce stress and make the mother feel more comfortable. Emotional comfort and support of the mother can positively affect breastfeeding performance. Reducing emotional stress can increase milk production and help the mother have a better breastfeeding experience.

For this reason, this study was planned to determine the effect of the emotional liberation technique on breastfeeding in women experiencing motherhood sadness.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily agrees to participate in the study,
* Experiencing motherhood blues
* Being over 18 years old

Exclusion Criteria:

* • Leaving the study at any time,

  * Having any obstacle to communication

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women
Enrollment: 64 (Actual)
Dates: Start 2024-03-16 (Actual); Primary Completion 2024-07-23 (Actual); Study Completion 2024-08-10 (Actual)

PRIMARY OUTCOMES:
The Effect of Emotional Freedom Technique on Breastfeeding in Women Experiencing Maternity Blues | Procedure 1: Preliminary tests will be carried out and then the 1st EFT session will be held. 2nd Procedure: After 10 days, the first final tests will be performed and then the second EFT session will be held.
  Emotional Freedom Technique

CONTACTS AND LOCATIONS:
Locations (1):
- Trakya University, Edirne, Turkey (Türkiye)